CLINICAL TRIAL: NCT04002596
Title: A Feasibility Study to Evaluate Safety and Initial Effectiveness of ExAblate Transcranial MR Guided Focused Ultrasound for Unilateral Thalamotomy in the Treatment of Medication-Refractory Tremor Dominant Idiopathic Parkinson's Disease
Brief Title: Safety and Initial Effectiveness of Transcranial MR Guided Focused Ultrasound for the Treatment of Parkinson's Disease
Acronym: TDPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD001J
Record Dates: First submitted 2019-01-07; First posted 2019-06-28 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: ExAblate Neuro Treatment Group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ExAblate MRgFUS treatment (Experimental): Ablation of Thalamus Vim nucleus with ExAblate 4000 Neuro MRgFUS for TDPD
  Interventions: Device: ExAblate Neuro Thalamotomy Treatment

INTERVENTIONS:
Device: ExAblate Neuro Thalamotomy Treatment — Non-invasive Focused Ultrasound Ablation of Thalamus Vim nucleus using ExAblate MRgFUS system for treatment Tremor Dominant Parkinson Disease
  Other Names: MRgFUS Vim ablation; Non-invasive Focused Ultrasound Ablation of Thalamus Vim nucleus

SUMMARY:
Safety and Effectiveness in ExAblate Neuro treatment of medication-refractory tremor in subjects with idiopathic Parkinson's disease.

DETAILED DESCRIPTION:
The goal of this prospective, single-arm, multi-site, feasibility study is to develop data to evaluate the safety and effectiveness of unilateral focused ultrasound thalamotomy using this ExAblate Transcranial System in the treatment of medication-refractory tremor resulting from idiopathic Parkinson's disease.

The Indications for Use claim for this system is: treatment of medication-refractory tremor in subjects with idiopathic Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, age 30 years and older
2. Subjects who are able and willing to give informed consent and able to attend all study visits through 3 Months
3. Subjects with a diagnosis of idiopathic PD as confirmed from clinical history and examination by a movement disorder neurologist at the site
4. All subjects included in this study will have a TD/PIGD ratio > 1.15 in the medicated [ON] state as calculated from the UPDRS formula as described by S, et. al., [74].

   Note: Ratios for TD/PIGD that are greater than or equal to 1.15 are defined as TDPD. PIGD includes those with a ratio of less than or equal to 0.9. Scores of greater than 0.9 and less than 1.15 are considered a mixed subtype.
5. Subject demonstrates a resting tremor severity score of greater than or equal to 3 in the hand/arm as measured by the medicated (ON) MDS-UPDRS question 3.17 or a postural/action tremor greater than or equal to a 2 for question 3.15 or 3.16.
6. Significant disability due to PD tremor despite medical treatment (CRST score of 2 or above in any one of the items 16-23 from the Disability subsection of the CRST: [speaking, feeding other than liquids, bringing liquids to mouth, hygiene, dressing, writing, working, and social activities])
7. Tremor remains disabling when medical therapy is optimal or not tolerated for the treatment of other cardinal signs of PD (bradykinesia, rigidity, etc), as determined by a movement disorders neurologist at the site
8. Subjects should be on a stable dose of all PD medications for 30 days prior to study entry.
9. The thalamus must be apparent on MRI such that targeting of the Vim nucleus can be performed indirectly by measurement from a line connecting the anterior and posterior commissures of the brain.
10. Subject is able to communicate sensations during the ExAblate Transcranial procedure.

Exclusion Criteria:

1. Subjects with unstable cardiac status including:

   1. Unstable angina pectoris on medication
   2. Subjects with documented myocardial infarction within six months of protocol entry
   3. Significant congestive heart failure defined with ejection fraction < 40
   4. Subjects with unstable ventricular arrhythmias
   5. Subjects with atrial arrhythmias that are not rate-controlled
2. Subjects exhibiting any behavior(s) consistent with ethanol or substance abuse as defined by the criteria outlined in the DSM-IV as manifested by one (or more) of the following occurring within the preceding 12 month period:

   1. Recurrent substance use resulting in a failure to fulfill major role obligations at work, school, or home (such as repeated absences or poor work performance related to substance use; substance-related absences, suspensions, or expulsions from school; or neglect of children or household).
   2. Recurrent substance use in situations in which it is physically hazardous (such as driving an automobile or operating a machine when impaired by substance use)
   3. Recurrent substance-related legal problems (such as arrests for substance related disorderly conduct)
   4. Continued substance use despite having persistent or recurrent social or interpersonal problems caused or exacerbated by the effects of the substance (for example, arguments with spouse about consequences of intoxication and physical fights).
3. Severe hypertension (diastolic BP > 100 on medication)
4. Subjects with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
5. Significant claustrophobia that cannot be managed with mild medication.
6. Current medical condition resulting in abnormal bleeding and/or coagulopathy
7. Patient with severely impaired renal function with estimated glomerular filtration rate <30 mL/min/1.73m2 (or per local standards should that be more restrictive) and/or who is on dialysis;
8. Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month of focused ultrasound procedure
9. Subjects with risk factors for intraoperative or postoperative bleeding as indicated by: platelet count less than 100,000 per cubic millimeter, a documented clinical coagulopathy, or INR coagulation studies exceeding the institution's laboratory standard
10. History of intracranial hemorrhage
11. History of multiple strokes, or a stroke within past 6 months
12. Subject who weigh more than the upper weight limit of the table or subjects who will not fit into the MR scanner
13. Subjects who are not able or willing to tolerate the required prolonged stationary supine position during treatment.
14. Are participating or have participated in another clinical trial in the last 30 days
15. Subjects unable to communicate with the investigator and staff.
16. Presence of central neurodegenerative disease, including but not limited to Parkinson-plus syndromes, suspected on neurological examination. These include: multisystem atrophy, progressive supranuclear palsy, corticobasal syndrome, dementia with Lewy bodies, and Alzheimer's disease.
17. Any suspicion that Parkinsonian symptoms are a side effect from neuroleptic medications.
18. Presence of significant cognitive impairment as determined with a score ≤ 24 on the Mini Mental Status Examination (MMSE)
19. Unstable psychiatric disease, defined as active uncontrolled depressive symptoms, psychosis, delusions, hallucinations, or suicidal ideation. Subjects with stable, chronic anxiety or depressive disorders may be included provided their medications have been stable for at least 60 days prior to study entry and if deemed appropriately managed by the site neuropsychologist
20. Subjects with significant depression as determined following a comprehensive assessment by a neuropsychologist. Significant depression is being defined quantitatively as a score of greater than 14 on the Beck Depression Inventory.
21. Legal incapacity or limited legal capacity as determined by the neuropsychologist
22. Subjects with a history of seizures within the past year
23. Subjects with brain tumors
24. Subjects with intracranial aneurysms requiring treatment or arterial venous malformations (AVMs) requiring treatment.
25. Any illness that in the investigator's opinion preclude participation in this study.
26. Pregnancy or lactation.
27. Subjects who have had deep brain stimulation or a prior stereotactic ablation of the basal ganglia
28. Subjects with remarkable atrophy and poor healing capacity of the scalp (> 30% of the skull area traversed by the sonication pathway) will be excluded from this study
29. Subjects who have an Overall Skull Density Ratio of 0.30 (±0.05) or less as calculated from the screening CT.

    * It should be noted that for those candidates whose SDR ratio score is within the standard deviation, full technical assessment should be performed and reviewed by study investigator with the support of the sponsor.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2019-09-04 (Actual)

PRIMARY OUTCOMES:
Clinical Rating Scale for Tremor | 3 Months after Treatment
  Primary effectiveness will be a comparison of the CRST scores at baseline vs. 3 months. (Range 0-152, scores are combined, the higher the score, the greater the clinical level of tremor, the worse clinical outcome is)
Severity of Device and Procedure related complications | 1 year
  To evaluate the incidence and severity of adverse events (AEs) associated with the ExAblate Transcranial thalamotomy of medication-refractory, tremor dominant PD after the ExAblate treatment and during the follow-up period of up up to 1 year

SECONDARY OUTCOMES:
Clinical Rating Scale for Tremor, Total Score | 1 year
  On-medication, total tremor (CRST) score (Range 0-152, scores are combined, the higher the score, the greater the clinical level of tremor, the worse clinical outcome is)
Clinical Rating Scale for Tremor, Part C | 1 year
  Level of disability measured from Part C subsection of CRST - Subcore of sections 16 to 23 (Range 0-32, scores are combined, the higher the scub-score, the greater the level of subject's disability, the worse clinical outcome is)
Parkinson's Disease Questionnaire - 39 | 1 year
  Quality of life assessment with PDQ-39 (Range 0-156, scores are combined, the higher the score, the greater the level of clinical expression of Parkinson Disease, the worse clinical outcome is)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Bernstein, Study Director — InSightec
Locations (1):
- Shonan Fujisawa Tokushukai Hospital, Fujisawa, Kanagawa, Japan

IPD SHARING:
Plan to Share IPD: No